CLINICAL TRIAL: NCT03017040
Title: In Vivo Kinematics of Scapolunate Interosseous Ligament Injuries
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough research staff
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Neal Chung-Jen Chen, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015P001271
Record Dates: First submitted 2016-12-07; First posted 2017-01-11 (Estimated); Results first posted 2018-09-17 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Scapholunate Ligament Tear
MeSH Terms: interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scapholunate tear (Experimental): Subjects with a full scapholunate tear will have a CT scan and fluoroscopy images taken
  Interventions: Device: CT scan; Device: Fluoroscopy Scan
- Control Wrist (Active Comparator): Subjects will have a CT scan and fluoroscopy image taken of the contralateral wrist serve as the control.
  Interventions: Device: CT scan; Device: Fluoroscopy Scan

INTERVENTIONS:
Device: CT scan — A CT scan of the wrist
Device: Fluoroscopy Scan — A fluoroscopy scan of the wrist.

SUMMARY:
The investigators hypothesize that there is no relationship between in vivo kinematic abnormalities and patient-rated outcomes for scapholunate interosseous ligament injuries (SLIL)

The secondary null hypotheses are that: There are no kinematic differences between subjects with unilateral, symptomatic, full thickness scapholunate ligament tears in comparison to the contralateral wrist without scapholunate ligament injury.

The investigators aim to answer to the below questions:

* What are baseline validated outcomes for subjects with SLIL injury?
* What are baseline physical measures (range of motion, Jamar Dynamometry)?

DETAILED DESCRIPTION:
In vivo kinematics of the normal wrist has been studied previously, but few studies have characterized the wrist with a SLIL injury. There are few studies evaluating validated patient-rated outcomes for patients with SLIL injury. The goal of this study would be to evaluate to what degree kinematic abnormalities affect patient-rated outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a unilateral full thickness scapholunate ligament tear diagnosed by radiographs or advanced imaging

Exclusion Criteria:

* Patients with a partial thickness scapholunate ligament tear
* Patients with radiographic arthrosis
* Patients with prior wrist injury
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Chen, MD, Principal Investigator — Massachusetts General Hospital

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Wrists
Groups:
- Scapholunate Tear: Subjects with a full scapholunate (SL) tear will have a CT scan and fluoroscopy images taken. Subjects will enroll the injured wrist into the SL tear group and uninjured wrist into the control group. Thus each participant will flow into both study arms/groups and may appear to be counted twice, however, for this study we focus on number of wrists.
  CT scan: A CT scan of the wrist
  Fluoroscopy Scan: A fluoroscopy scan of the wrist.
- Control Wrist: Subjects will have a CT scan and fluoroscopy image taken of the contralateral wrist serve as the control. Subjects will enroll the injured wrist into the SL tear group and uninjured wrist into the control group. Thus each participant will flow into both study arms/groups and may appear to be counted twice, however, for this study we focus on number of wrists.
  CT scan: A CT scan of the wrist
  Fluoroscopy Scan: A fluoroscopy scan of the wrist.
Period: Overall Study
Arm/Group | Scapholunate Tear | Control Wrist
Started | 1; 1 Wrists (Participants enroll one wrist into each group,thus, one participant flows into both groups.) | 1; 1 Wrists (Participants enroll one wrist into each group,thus, one participant flows into both groups.)
Completed | 0; 0 Wrists | 0; 0 Wrists
Not Completed | 1; 1 Wrists | 1; 1 Wrists

BASELINE CHARACTERISTICS:
Population: One subject accounts for scapholunate tear and control wrist, i.e., one subject enrolled for two study wrists.
Groups:
- Participants With Unilateral Scapholunate Tear: All subjects with a full scapholunate (SL) tear will have a CT scan and fluoroscopy images taken. The injured wrist will enroll in the SL tear group and the uninjured wrist as the control wrist.
  CT scan: A CT scan of the wrist
  Fluoroscopy Scan: A fluoroscopy scan of the wrist.
Arm/Group | Participants With Unilateral Scapholunate Tear
Number analyzed (Participants) | 1
Age, Continuous [Mean (Full Range); unit: years] | 47 [47 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Patient Rated Wrist Evaluation (PRWE)
Description: The questionnaire will help the investigators determine how much difficulty the subject has had with the injured wrist in the past week.
Time Frame: at enrollment
Population: The paper-based questionnaire was not scored and tallied, thus not analyzed.
Arm/Group | Scapholunate Tear | Control Wrist
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: SF-12 Patient Questionnaire
Description: The SF-12 questionnaire will help the investigators determine how well subjects are able to do usual activities
Time Frame: at enrollment
Population: The paper-based questionnaire was not scored and tallied, thus not analyzed.
Arm/Group | Scapholunate Tear | Control Wrist
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: DASH Questionnaire
Description: The DASH questionnaire will help the investigators determine the level of disability subjects face from the wrist injury.
Time Frame: at enrollment
Population: The paper-based questionnaire was not scored and tallied, thus not analyzed.
Arm/Group | Scapholunate Tear | Control Wrist
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Scapholunate Tear | Control Wrist
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT03017040/Prot_SAP_000.pdf